CLINICAL TRIAL: NCT06459102
Title: The Effect of Motor Learning Exercises on Motor Imagery, Function, Pain and Grip Strength in Individuals With Chronic Lateral Epicondylitis
Brief Title: The Effect of Motor Learning Exercises on Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KaratayUH12
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2024-06

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Learning (Experimental): In addition to the conventional physiotherapy program, motor learning exercise will be performed for 6 weeks, 3 sessions per week. For the exercise, the participant will sit in a chair with back support, in front of a table, with arms on the table. The participant will wear a glove with an IMU sensor on the upper surface and a pressure sensor on the palm, and a cylinder will be placed in the palm. The participant will be asked to bring the wrist into extension and then back into flexion while grasping the cylinder with maximum force. The participant will be asked to maintain maximum strength during the entire movement. The participant will be given visual feedback on muscle strength and range of motion of the wrist on the monitor in front of them throughout the movement. The same protocol will be applied by keeping the size of the cylinder in the participant's palm the same and changing the weight.
  Interventions: Other: Motor Learning
- Control (Active Comparator): The control group will receive a conventional physiotherapy program for 4 weeks, 5 days a week. Eccentric training for the extensor carpi radialis brevis (ECRB) muscle, the most affected wrist extensor tendon, and static stretching exercises for the ECRB muscle will be given. For eccentric training, the weight that the patients can lift in 10 maximal repetitions will be calculated and they will be asked to work with this weight. The best stretching position for the ECRB tendon is extension of the elbow joint, pronation of the forearm and flexion of the wrist with ulnar deviation. Each participant will be taught to perform each exercise for 10 repetitions and 10 seconds. Patients will perform these exercises in a sitting position. In the control group, daily exercises will be performed under the supervision of a physiotherapist.
  Interventions: Other: Control

INTERVENTIONS:
Other: Motor Learning — In addition to the conventional physiotherapy program .... per week for 4 weeks Sessions of motor learning exercise will be performed. For the exercise, the participant will sit in a chair with back support, in front of a table, with arms on the table. The participant will wear a glove with an IMU sensor on the upper surface and a pressure sensor on the palm, and a cylinder will be placed in the palm. The participant will be asked to bring the wrist into extension and then back into flexion while grasping the cylinder with maximum force. The participant will be asked to maintain maximum strength during the entire movement. The participant will be given visual feedback on muscle strength and range of motion of the wrist on the monitor in front of them throughout the movement. The same protocol will be applied by keeping the size of the cylinder in the participant's palm the same and changing the weight.
  Arms: Motor Learning
Other: Control — The control group will receive a conventional physiotherapy program for 4 weeks, 5 days a week. Eccentric training for the extensor carpi radialis brevis (ECRB) muscle, the most affected wrist extensor tendon, and static stretching exercises for the ECRB muscle will be given. For eccentric training, the weight that the patients can lift in 10 maximal repetitions will be calculated and they will be asked to work with this weight. The best stretching position for the ECRB tendon is extension of the elbow joint, pronation of the forearm and flexion of the wrist with ulnar deviation. Each participant will be taught to perform each exercise for 10 repetitions and 10 seconds. Patients will perform these exercises in a sitting position. In the control group, daily exercises will be performed under the supervision of a physiotherapist
  Arms: Control

SUMMARY:
The aim of this study was to determine the effect of motor learning training in addition to a 6-week conventional physiotherapy program on motor imagery, function pain and grip strength in individuals with chronic lateral epicondylitis. At the end of the study, it is aimed to develop a system for motor learning training in individuals with chronic lateral epicondylitis and to create a new exercise protocol.

DETAILED DESCRIPTION:
The study will include 46 volunteers aged 18-65 years. Participants will be randomly assigned to the Motor learning (n=23) and control (n=23) groups according to an internet-based randomization program.

The system to be used in the first phase of the study will be developed. The system will consist of a glove with a pressure sensor on the inner surface and an M-IMU sensor on the outer surface, a computer and a monitor. The pressure sensor on the inner surface will collect instantaneous data on grip force and the M-IMU sensor on the outer surface will collect instantaneous data on wrist movement. The software to be developed will process the instantaneous information from the sensors and reflect it to the monitor.

In the second phase of the study, the effectiveness of the motor learning exercise protocol to be applied with the developed system will be evaluated.

The motor learning group will receive 3 sessions of motor learning exercise per week for 6 weeks, 5 days a week, in addition to the conventional physiotherapy program.

The control group will receive eccentric training for the extensor carpi radialis brevis (ECRB) muscle and static stretching exercises for the ECRB muscle in addition to the conventional physiotherapy program 5 days a week for 6 weeks.

All evaluations of the participants will be performed blindly by an independent investigator before and at the end of the study.

Participants' motor imagery will be assessed through a left/right judgment task in which they must recognize whether hand images correspond to their left or right side using the Recognise™ application (Neuro Orthopaedic Institute, Adelaide, Australia).

Participants' function will be assessed using the Patient Rated Tennis Elbow Evaluation (PRTEE), pain will be assessed using a visual analog scale, and grip strength will be assessed using a hydraulic hand dynamometer.

Activities of Daily Living The DASH questionnaire is a questionnaire that asks about physical activities and symptoms of disease. It helps to assess problematic arm, shoulder and hand activities. It is a 30-item questionnaire that assesses the patient's ability to perform certain upper limb activities. These activities include activities performed at home, whether there are complaints such as pain, weakness, tingling in the hand, arm or shoulder, sports activities, etc. The DASH is a self-report questionnaire in which patients can rate difficulties and interventions in their daily lives on a 5-point Likert scale. The lower the calculated DASH score, the better the patient's functionality.

Satisfaction Participants' satisfaction will be assessed through a satisfaction survey on technological rehabilitation practices.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of chronic LET by a physician and
* a pain score > 3 on the visual analog scale (VAS)

Exclusion Criteria:

* concomitant disorders of the wrist and forearm, such as elbow fracture or dislocation, and
* treatment with corticosteroid injections within the previous 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Motor imagery | Baseline, 6 weeks
  Motor imagery will be assessed through a left/right judgment task in which participants will need to recognize whether hand images correspond to their left or right side using the Recognise™ application (Neuro Orthopaedic Institute, Adelaide, Australia).

SECONDARY OUTCOMES:
Function | Baseline, 6 weeks
  Total scores range from 0 to 100, with higher scores indicating increased pain and loss of function
Elbow Pain | Baseline, 6 weeks
  Participants' pain will be assessed with a 10 cm visual analog scale. For pain, 0 (baseline) means no pain and the other end (10, endpoint) means very severe pain; the patient marks his/her pain level on this 10 cm line. The assessment will be done at night, at rest and patient activity pain.
Grip strength | Baseline, 6 weeks
  The maximal grip strength of the patients will be measured with a hydraulic hand dynamometer. Measurements will be performed in two positions. In the sitting position, measurements will be made in shoulder adduction, elbow 90 flexion, forearm neutral position, wrist 0-30 extension and 0-15 ulnar deviation. In standing position, shoulder abduction, elbow extension and forearm neutral position will be measured. Patients will be asked to press the dynamometer with maximum force for 3 seconds and this value will be recorded as the maximum grip force. The measurements will be repeated three times at 30-second intervals on the affected limb and the average of the measurements will be recorded.
Activities of Daily Living | Baseline, 6 weeks
  The DASH questionnaire is a questionnaire that asks about physical activities and symptoms of disease. It helps to assess problematic arm, shoulder and hand activities. It is a 30-item questionnaire that assesses the patient's ability to perform certain upper limb activities. These activities include activities performed at home, whether there are complaints such as pain, weakness, tingling in the hand, arm or shoulder, sports activities, etc. The DASH is a self-report questionnaire in which patients can rate difficulties and interventions in their daily lives on a 5-point Likert scale. The lower the calculated DASH score, the better the patient's functionality.
Treatment satisfaction | Baseline, 6 weeks
  Participants' satisfaction will be assessed through a satisfaction survey on technological rehabilitation practices

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gercek H, Cihan E, Celik F, Sonmez Unuvar B, Sari Z. Pain, grip strength, and motor imagery reaction time are associated with pain and disability in individuals with chronic lateral elbow tendinopathy. Musculoskelet Sci Pract. 2026 Feb;81:103463. doi: 10.1016/j.msksp.2025.103463. Epub 2025 Dec 1. PMID 41349351